CLINICAL TRIAL: NCT00764023
Title: A Multi-Center Protocol for Obtaining and Storing Human Samples for Immediate or Future Microbial, Immune,or Host-Microbe Scientific Study
Brief Title: A Multi-Center Protocol for Obtaining and Storing Human Samples for Immediate or Future Microbial, Immune, or Host-Microbe Scientific Study
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Prinicipal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-010
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Infections
Keywords: wound debridement; removed orthopedic implants; removed catheters or shunts; excised tonsils, amputated tissue; sputum; stool; other excretions.
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The intent of this protocol is to salvage human-related material that is normally destined for destruction, so it can be used in infection-related scientific studies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- No treatment
- human samples

SUMMARY:
The intent of this protocol is to salvage human-related material that is normally destined for destruction, so it can be used in infection-related scientific studies. This clinical material can be studied in order to better understand the molecular, cellular, or ecological components of the infected or potentially infected tissue or device.

DETAILED DESCRIPTION:
The samples can include material such as wound debridement, removed orthopedic implants, removed catheters or shunts, excised tonsils, amputated tissue, sputum, stool, or other excretions. The samples can be cultured for microbes, examined using microscopy, or analyzed using molecular techniques. The studies can examine microbes or the host's response to microbes by examining the nucleic acids (e.g. 16S DNA, mRNA), proteins, or other metabolites.

ELIGIBILITY:
Inclusion Criteria:

1. The Subject must be 18 years of age or older
2. The Subject must be mentally competent as determined by the Investigator, or have a Legally Authorized Representative.

Exclusion Criteria:

1. The Subject may not be currently incarcerated.
2. The Subject may not be knowingly pregnant.
3. The Subject may not be institutionalized.
4. The Subject may not be an employee or student of the investigator or sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The samples can include material such as wound debridement, removed orthopedic implants, removed catheters or shunts, excised tonsils, amputated tissue, sputum, stool, or other excretions.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2008-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The samples can be cultured for microbes, examined using microscopy, or analyzed using molecular techniques. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Randall Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States

REFERENCES:
- [Result] A Possible Role of Bacterial Biofilm in the Pathogenesis of Atherosclerosis Bacteriol Parasitol Volume 3 • Issue 1 • 1000127 ISSN:2155-9597 JBP an open access journal